CLINICAL TRIAL: NCT06561607
Title: A Randomized, Open, Parallel-Controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of TQB2102 for Injection Versus Investigator-Selected Chemotherapy in HER2 Low-Expressing Recurrent/Metastatic Breast Cancer
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of TQB2102 for Injection Versus Investigator-Selected Chemotherapy in HER2 Low-Expressing Recurrent/Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-III-01
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2102 for Injection (Experimental): Administered by intravenous drip, 7.5 mg/kg per dose, 21 days as a treatment cycle.
  Interventions: Drug: TQB2102 for Injection
- Chemotherapy drug (Capecitabine/Paclitaxel/Albumin Paclitaxel) (Active Comparator): Based on each patient's condition and previous treatment history, the investigator will select one of the following chemotherapy drugs for treatment.
  * Capecitabine
  * Paclitaxel
  * Albumin Paclitaxel
  Interventions: Drug: Chemotherapy drug (Capecitabine/Paclitaxel/Albumin Paclitaxel)

INTERVENTIONS:
Drug: TQB2102 for Injection — TQB2102 is a next-generation HER2 Antibody-Drug Conjugate (ADC) drug proposed for patients with HER2 low-expressing breast cancer.
  Arms: TQB2102 for Injection
Drug: Chemotherapy drug (Capecitabine/Paclitaxel/Albumin Paclitaxel) — Based on each patient's condition and previous treatment history, the investigator will select one of the chemotherapy drugs for treatment.
  * Capecitabine: 1000-1250 mg/m2 twice daily, administered consecutively on day 1-14, 21 days as a treatment cycle.
  * Paclitaxel: 175 mg/m2, IV infusion, administered Day1 per cycle, 21 days as a treatment cycle. OR 80 mg/m2 by IV infusion administered weekly.
  * Albumin Paclitaxel: 260 mg/m2, IV infusion, administered every cycle of Day1 for 21 days as a treatment cycle. 100 mg/m2 or 125 mg/m2, IV infusion, administered every cycle of Day 1 and Day 8 for 21 days as a treatment cycle; or Day 1, Day 8, and Day 15 administered every cycle for 28 days as a treatment cycle.
  Arms: Chemotherapy drug (Capecitabine/Paclitaxel/Albumin Paclitaxel)

SUMMARY:
The study is a Phase III, randomized, multicenter, open-label study in HER2-low, HR+ metastatic breast cancer subjects who are patients with locally advanced or metastatic breast cancer with low HER2 expression in the recurrent metastatic stage who have not received chemotherapy. The primary objective of the study is to determine the efficacy and safety of TQB2102 compared to investigator-selected single-agent chemotherapy in the target population. 542 subjects with HER2 immunohistochemistry (IHC )2+/ in situ hybridization (ISH)- and IHC 1+ (HER2-low) expression will be enrolled in 1:1 randomized groups to receive TQB2102 or investigator's choice of single-agent chemotherapy (capecitabine, paclitaxel, or albumin-paclitaxel) until progression of disease (PD), as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1. 1, unless there are unacceptable toxicity, withdrawal of consent, or meeting other discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily enrolled in this study with good compliance;
* Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-1;
* Pathologically confirmed locally advanced or metastatic breast cancer with low HER2 expression and unresectable:
* Defined hormone receptor (HR) status.
* Imaging-confirmed disease progression (during or after completion of the most recent treatment);
* Have at least one measurable lesion according to RECIST 1.1 criteria;
* Good major organ function.

Exclusion Criteria:

* The presence or current concurrent presence of other malignant tumors within 5 years prior to randomization. ;
* Unresolved toxic reactions above Common Terminology Criteria for Adverse Events (CTC AE) grade 1 due to any prior therapy;
* Major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of the pre-randomization period;
* Prolonged unhealed wounds or fractures;
* Previous history of interstitial lung disease/pneumonia requiring steroidal drug intervention;
* The presence of moderate to severe pulmonary dysfunction/disease within 3 months prior to randomization;
* The presence of an arterial/deep vein thrombotic event within 6 months prior to randomization;
* The presence of a medical condition that interferes with intravenous administration, intravenous blood collection, or inability to swallow, chronic diarrhea, intestinal obstruction, or the presence of other factors that interfere with the administration and absorption of medications;
* The presence of grade ≥2 myocardial ischemia or myocardial infarction, cardiac arrhythmias (including QT corrected (QTc) ≥450ms (men) and QTc ≥470ms (women)) and grade ≥2 congestive heart failure (New York Heart Association (NYHA) classification); angina pectoris requiring antianginal medication; and clinically significant heart valve disease;
* Active or uncontrolled ≥ CTC AE grade 2 infection present within 14 days prior to randomization;
* Cirrhosis of the liver, active hepatitis that is not well controlled;
* Renal failure requiring hemodialysis or peritoneal dialysis;
* History of immunodeficiency, including HIV-positive or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
* Those with routine urinalysis suggestive of urinary protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g;
* Those who have used immunosuppressive or systemic hormone therapy for immunosuppression within 2 weeks prior to randomization;
* Those with a history of psychotropic substance abuse that cannot be abstained from or those with psychiatric disorders;
* Tumor-related symptoms and treatments:

  1. Subjects who have been treated with other antineoplastic agents such as chemotherapy, radical radiotherapy, or immunotherapy within 4 weeks prior to randomization, or who are still within 5 half-lives of the drug (whichever occurs shortest);
  2. Treatment with endocrine therapy, molecularly targeted therapy, or a proprietary Chinese medicine with an anti-tumor indication as specified in the National Medical Products Administration (NMPA) approved drug insert within 2 weeks prior to randomization;
  3. Presence of carcinomatous lymphadenitis, or uncontrollable pleural effusion, ascites, and pericardial effusion of moderate volume or greater that requires repeated drainage to relieve clinical symptoms, or who have received drainage of plasmapheresis for therapeutic purposes within 2 weeks prior to randomization;
  4. Known carcinomatous meningitis or clinically active central nervous system metastases;
  5. Severe bone damage resulting from tumor bone metastases;
* Those who have received a control chemotherapeutic agent of the investigator's choice during the recurrent metastatic phase or for whom a control chemotherapeutic agent of the investigator's choice is inappropriate for reasons such as intolerance or contraindication to that agent;
* Has received prior anti-HER2 therapy;
* Who have developed hypersensitivity to humanized monoclonal antibody products;
* Those who have developed an allergy to any of the study drugs or any component or excipient in the drugs;
* Who have participated in and used another antitumor clinical trial drug within 4 weeks prior to randomization;
* Subjects who, in the judgment of the investigator, have a concomitant disease that seriously jeopardizes the safety of the subject or interferes with the completion of the study, or who are deemed to have other reasons for being unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in subjects with HR-positive, HER2 low-expressing recurrent/metastatic breast cancer as assessed by Independent Review Committee (IRC) | Up to 25 months
  Designed to demonstrate that in subjects with HR-positive, HER2 low-expressing recurrent/metastatic breast cancer, TQB2102 for injection significantly prolongs progression-free survival in subjects compared to investigator-selected chemotherapy.

SECONDARY OUTCOMES:
Progression-free survival (PFS) in subjects with HER2 low-expressing recurrent/metastatic breast cancer as assessed by IRC | Up to 25 months
  Designed to demonstrate that in subjects with HER2 low-expressing recurrent/metastatic breast cancer, TQB2102 for injection significantly prolongs progression-free survival in subjects compared to investigator-selected chemotherapy.
Progression-free survival (PFS) as assessed by investigators in the HR-positive, HER2 low-expressing population | Up to 25 months
  To evaluate progression-free survival (PFS) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HR-positive, HER2 low-expressing recurrent/metastatic breast cancer.
Investigator-assessed overall survival (OS) in HR-positive, low HER2-expressing population. | Up to 25 months
  To evaluate the overall survival (OS) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HR-positive, HER2 low-expressing recurrent/metastatic breast cancer.
Overall survival (OS) as assessed by investigators in the HR-positive, HER2 low-expressing population | Up to 25 months
  To evaluate the objective remission rate (ORR) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HR-positive, HER2 low-expressing recurrent/metastatic breast cancer.
Duration of remission (DOR) as assessed by investigators in the HR-positive, HER2 low-expressing population | Up to 25 months
  To evaluate the duration of remission (DOR) of injectable TQB2102 compared to investigator-selected chemotherapy in subjects with HR-positive, HER2 low-expressing recurrent/metastatic breast cancer.
Investigator-assessed clinical benefit rate (CBR) in the HR-positive, low HER2-expressing population | Up to 25 months
  To evaluate the clinical benefit rate (CBR) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HR-positive, HER2 low-expressing recurrent/metastatic breast cancer.
Progression-free survival (PFS) as assessed by investigators in the HER2 low expression population | Up to 25 months
  To evaluate progression-free survival (PFS) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
Overall survival (OS) as assessed by investigators in the HER2 low expression population | Up to 25 months
  To evaluate the overall survival (OS) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
Duration of remission (DOR) as assessed by investigators in the HER2 low expression population | Up to 25 months
  To evaluate the duration of remission (DOR) of injectable TQB2102 compared to investigator-selected chemotherapy in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
Objective remission rate (ORR) as assessed by investigators in the HER2 low expression population | Up to 25 months
  To evaluate the objective remission rate (ORR) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
Clinical benefit rate (CBR) as assessed by investigators in the HER2 low expression population | Up to 25 months
  To evaluate the clinical benefit rate (CBR) of TQB2102 for injection versus investigator-selected chemotherapy in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and indicators of abnormal laboratory tests | Up to 52 months
  To evaluate the safety of TQB2102 for Injection compared to investigator-selected chemotherapy in subjects with HER2 low-expressing recurrent/metastatic breast cancer, including: the incidence and severity of adverse events (AEs), abnormal laboratory test values, and serious adverse events (SAEs).
Blood concentrations of the ADC drug TQB2102, total antibodies, and the small molecule toxin TQ22723 | Within 1 hour prior to the start of infusion for Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 7, and Cycle 12, and 0.5 to 2 hours after the end of infusion for Cycle 2, Cycle 3, Cycle 4, Cycle 7, and Cycle 12 (21 days as a treatment cycle).
  To evaluate the pharmacokinetic (PK) profile of TQB2102 for injection in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
  Within 1 hour prior to the start of infusion for Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 7, and Cycle 12, and 0.5 to 2 hours after the end of infusion for Cycle 2, Cycle 3, Cycle 4, Cycle 7, and Cycle 12 .
Immunogenicity of TQB2102: ADA incidence | Prior to (-60 min) the first day of dosing in Cycle 1, Cycle 2, Cycle 4, Cycle 7, and Cycle 12 (21 days as a treatment cycle), and at follow-up 30 days (±7 days) after the last dosing.
  To evaluate the immunogenicity (ADA) of TQB2102 for injection in subjects with HER2 low expression recurrent/metastatic breast cancer.

CONTACTS AND LOCATIONS:
Locations (34):
- China (34):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - AnHui Province Hospital West District, Hefei, Anhui
  - The first Affiliated hospital of anhui medical university, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University 2nd Affiliated Hospital, Quanzhou, Fujian
  - Zhangzhou Hospital in Fujian Province, Zhangzhou, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Sun Yet-Sen University Cancer Certer, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Guigang City People'S Hospital, Guigang, Guangxi
  - Cancer Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - The First affiliated hospital of GuangXi medical university, Nanning, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University Co., LTD, Guiyang, Guizhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - Hainan General Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Chengde Central Hospital, Chengde, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - Henan Cancar Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Hennan
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - The Second Hospital of DALIAN Medical University, Dalian, Liaoning
  - Binzhou Medical College Affiliated Hospital, Binzhou, Shandong
  - Binzhou People's Hospital, Binzhou, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Affiliated Hospital of North Scichuan Medical College, Nanchong, Sichuan
  - Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang